CLINICAL TRIAL: NCT05632107
Title: Comparison of an Acceleromyography- and Electromyography-based Neuromuscular Monitor With TOF-Watch ® Monitor：a Pilot Study
Brief Title: Comparison of an Acceleromyography- and Electromyography-based Neuromuscular Monitor With TOF-Watch ® Monitor
Status: Recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hua Zheng, Associate Professor, Huazhong University of Science and Technology
Other Study IDs: TJMZK202201
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Neuromuscular Blockade
Keywords: neuromuscular blocking agents; residual neuromuscular blockade; neuromuscular monitoring; acceleromyography; electromyography
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TOF-Watch®；DELSYS® Wireless surface EMG — TOF-Watch® is the most widely accepted AMG-based neuromuscular monitor; and DELSYS® Wireless surface EMG is a new technology that allows for the simultaneous acquisition of EMG and AMG signals in a wireless manner.

SUMMARY:
A quantitative neuromuscular monitoring device is desirable to titrate the depth of neuromuscular block (NMB) during a procedure, and to prevent residual effects after removal of the endotracheal tube. Unfortunately, the most widely used monitoring technique acceleromyography (AMG) typically implies a series of cumbersome installation and calibration procedures that frequently precludes correct use of these devices in clinical practice. Electromyography (EMG) has recently attracted a lot of attention as an alternative strategy to compensate for the deficiency of AMG-based neuromuscular monitors. Nowadays, a new technology that allows for the simultaneous acquisition of EMG and AMG signals is commercially available. Although its reliability has been rapidly accepted in Physical Medicine and Rehabilitation, the use of the technique in neuromuscular monitoring has never been reported. The aim of the present study is to assess the validity of the new device for estimating the neuromuscular block by comparing with TOF Watch®-SX, which is the most widely accepted AMG-based neuromuscular monitor that has been practiced in the clinical arena for decades.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 18 yr
* American Society of Anesthesiologists Physical Status I to III
* Elective surgery requiring muscle relaxation
* Patients participated voluntarily and signed informed consent

Exclusion Criteria:

* Patients with known neuromuscular disorder
* Stroke
* Patients with a history of allergic reaction toneuromuscular blocking agents
* Use of medications that might interfere with neuromuscular transmission
* Any previous injury to the examined arm that might influence nerve conduction parameters
* Pacemaker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need to be treated surgically under general anesthesia and are going to receive neuromuscular blocking agents.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessing the correlation between the train-of-four (TOF) obtained from the 2 devices | Perioperative data
Assessing the correlation between the posttetanic count (PTC) obtained from the 2 devices | Perioperative data

SECONDARY OUTCOMES:
Screening for eligible individual signal sources from the multiplex information of the new technology for improving neuromuscular monitoring | Perioperative data

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zheng, Dr., Study Director — Department of Anesthesiology, Tongji Hospital
Locations (2):
- China (2):
  - Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei